CLINICAL TRIAL: NCT05764577
Title: Intraabdominal Pressure Increases Peri-operatively in Patients Undergoing DIEP Flap Reconstruction: A Prospective Study Linking High IAP to Non-fatal Lung Embolism in One Patient
Brief Title: DIEP Flap Surgery and Intraabdominal Pressure
Status: Completed | Type: Observational
Sponsor: Aalborg University Hospital (Other)
Responsible Party: Principal Investigator, Nikolaj Warming, Principal investigator, Aalborg University Hospital
Other Study IDs: 2021-082
Record Dates: First submitted 2023-02-23; First posted 2023-03-10 (Actual); Last update posted 2023-03-10 (Actual); Status verified 2023-03

CONDITIONS: Intraabdominal Hypertension; Breast Neoplasms
MeSH Terms: conditions — Intra-Abdominal Hypertension; Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Surgical intervention: Participants who underwent secondary DIEP flap breast reconstruction
  Interventions: Procedure: DIEP flap surgery

INTERVENTIONS:
Procedure: DIEP flap surgery — Removal off the DIEP flap followed by closure of the rectus sheath and abdominal skin.

SUMMARY:
Aim: The primary aim of this study is to test if closure of the abdominal donor site increases the Intraabdominal Pressure (IAP) in women undergoing secondary Deep Inferior epigastric perforator (DIEP) flap breast reconstruction.

Materials and method: By an Unometer, attached to a standard catheter in the bladder, we measured the intravesical pressure as a surrogate marker for the IAP, at baseline, immediate after- and 24 hours after abdominal skin closure, for 13 patients.

ELIGIBILITY:
Inclusion Criteria:

* Females undergoing secondary DIEP flap breast reconstruction.
* Performance status 1-2

Exclusion Criteria:

* Performance status above 2.
* Untreated hypertension or atrial fibrillation

Performance status evalutated using American Society of Anaesthesiologists' (ASA) classification of Physical Health.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: Females undergoing secondary DIEP flap breast reconstruction. Performance status ASA 1-2
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2021-04-19 (Actual); Primary Completion 2021-11-29 (Actual); Study Completion 2022-01-25 (Actual)

PRIMARY OUTCOMES:
Changes from Baseline in intraabdominal pressure at timepoint immediate after- and 24 hours after abdominal skin closure. | Baseline, immediate after- and 24 hours after abdominal skin closure
  : By an Unometer, attached to a standard catheter in the bladder, we measured the intravesical pressure as a surrogate marker for the IAP, at baseline, immediate after- and 24 hours after abdominal skin closure

CONTACTS AND LOCATIONS:
Locations (1):
- University hospital Aalborg, Aalborg, North Jutland, Denmark

IPD SHARING:
Plan to Share IPD: Undecided